CLINICAL TRIAL: NCT07232784
Title: Serial Measurement of Pancreatic Stone Protein (PSP) for the Early Recognition and Diagnosis of Sepsis in Intensive Care Unit (ICU) Patients in China: A Multicenter, Prospective, Biomarker-result-blinded Observational Study
Brief Title: Serial Measurement of Pancreatic Stone Protein (PSP) for Sepsis Early Detection in ICU Patients
Status: Completed | Type: Observational
Sponsor: Fapon Biotech Inc. (Industry)
Collaborators: Shenzhen People's Hospital (Other); Shenzhen Third People's Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); ZhuHai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fapon-IIT-PSP-01; IIT-PSP-01 (Other: Fapon Biotech)
Record Dates: First submitted 2025-09-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Adult Patients at High Risk of Sepsis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Blood Sampling (whole blood and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients at high risk of sepsis presenting to Intensive Care Units (ICUs) and Emergency: Adult patients at high risk of sepsis presenting to Intensive Care Units (ICUs) and Emergency, who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled in the trial and collected 3 ml of peripheral venous blood samples daily (together with blood tests such as complete blood count for normal diagnosis and treatment purposes) until the diagnosis of sepsis or other diseases was confirmed, for central analysis of biomarkers of inflammation, infection and/or sepsis, including but not limited to Pancreatic Stone Protein [① PSP (CLIA, Fapon Biotech); ② EU IVDR-marked IVD PSP capsule on the point-of-care abioSCOPE® device (Abionic SA)], C-reactive protein (CRP), Procalcitonin (PCT), etc.
  Interventions: Device: blood sampling

INTERVENTIONS:
Device: blood sampling — Subjects will be collected 3 ml of peripheral venous blood samples daily (together with blood tests such as complete blood count for normal diagnosis and treatment purposes) until the diagnosis of sepsis or other diseases was confirmed, for central analysis of biomarkers of inflammation, infection and/or sepsis, including but not limited to Pancreatic Stone Protein [① PSP (CLIA, Fapon Biotech); ② EU IVDR-marked IVD PSP capsule on the point-of-care abioSCOPE® device (Abionic SA)], C-reactive protein (CRP), Procalcitonin (PCT), Interleukin-6 (IL-6), Pro-Brain Natriuretic Peptide (pro-BNP), High-sensitivity cardiac troponin I (hs-cTnI), Serum amyloid A (SAA), Cystatin C (Cys C), Calprotectin (CAL), etc.

SUMMARY:
In this study, 250 patients with high-risk of sepsis will be enrolled, including ≥ 50 subjects with confirmed sepsis. Diagnostic criteria for sepsis should meet the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3), i.e., simultaneously meet the following two conditions: a) confirmed or suspected infection; b) the SOFA score has increased by ≥ 2 points compared with the baseline. Subjects who meet the inclusion criteria and do not meet the exclusion criteria will be collected 3 ml of peripheral venous blood samples daily (together with blood tests such as complete blood count for normal diagnosis and treatment purposes) until the diagnosis of sepsis or other diseases was confirmed.

During the blood collection period, relevant clinical information, laboratory examination results, treatment information and SOFA scores of the subjects will be collected. This study does not produce any intervention in the normal clinical diagnosis and treatment of the subjects. After the subjects were diagnosed with sepsis, a 28-day follow-up will be performed to record the number of days of ICU treatment and the survival of the subjects 7 and 28 days after the diagnosis of sepsis. If the subjects were diagnosed with septic shock during the follow-up period, they will be recorded as "Ds". If the subjects were still hospitalized in the study center, 3 ml of peripheral venous blood samples will be collected. The completion of the 28-day follow-up will be considered the end of the study.

This study aims to:

1. Comparing to reference method, the clinical diagnosis of sepsis (sepsis-3), and reference reagents, CE-marked IVD PSP capsule on the point-of-care abioSCOPE® device (Abionic SA), C-reactive protein (CRP) assay kit, procalcitonin (PCT) assay kit, etc., to verify and evaluate the comprehensive performance of PSP as a biomarker in the early recognition and diagnosis of sepsis manifesting within the first 3 days after testing. Diagnostic accuracy analysis [including sensitivity, specificity, positive predicted value, negative predicted value, positive likelihood ratio, negative likelihood ratio, area under ROC curve (AUC), etc.], and consistency analysis (including positive coincidence rate, negative coincidence rate, total coincidence rate, Kappa value, etc.) will be performed.

   1. The clinical performance of PSP for the diagnosis of sepsis will be evaluated based on the cross-sectional study data (on the day of confirmed visit).
   2. The clinical performance of PSP for recognition of sepsis manifesting within the first 3 days after testing will be evaluated based on the longitudinal study data (multiple visits data).
2. Comparing to the reference method and the reference reagent test results, try to use machine learning & deep learning methods to select a subset of relevant features (variable screening) from clinical information and biomarker data (CRP, PCT, IL-6, NT-proBNP, hs-cTnI, SAA, Cys C, CAL, etc.), to construct an innovative combined diagnostic model with PSP, "PSP+ X" model. The comprehensive performance of "PSP+X" model for the early recognition and diagnosis of sepsis manifesting within the first 3 days after testing will be evaluated. Diagnostic

   1. The clinical performance of "PSP+X" mode for the diagnosis of sepsis will be evaluated based on the cross-sectional study data (on the day of confirmed visit).
   2. The clinical performance of "PSP+X" mode for early recognition of sepsis manifesting within the first 3 days after testing will be evaluated based on the longitudinal study data (multiple visits data).

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients over 18 years old；
2. Patients at high risk of sepsis in any of the following:

   1. History of recent surgery or invasive medical procedures;
   2. Pneumonia, complicated urinary tract infections, abdominal infections, central nervous system infections, etc.;
   3. Severe trauma: such as the percentage of total body surface area (TBSA) burned > 15%, or serious traffic accident injuries, etc.;
3. Expected ICU stay for more than 4 days；
4. Have provided written informed consent or consent is given by the patient's legally designated representative.

Exclusion Criteria:

1. Patients diagnosed with sepsis;
2. Patients expected to die within 48 hours of admission to ICU；
3. Pregnancy；
4. Patient suffering from or known acute or chronic pancreatitis, pancreatic cancer or admitted after pancreatectomy; but if a patient develops any pancreatic disease during the ICU stay, he/she will remain in the study；
5. Patients with SOFA score < 2 but who have undergone blood purification;
6. Unable or unwilling to provide the required blood sample for testing；
7. Patients with unclear medical record information;
8. Patients with mental disorders and other disorders who cannot correctly understand informed consent;
9. Patients who subjectively refused to be enrolled in the study or who were judged not to be enrolled by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU admitted patients at high-risk of developing sepsis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of PSP to aid in the early recognition and diagnosis of sepsis manifesting within the first 3 days after testing | 1) Blood sample collection period: from enrollment to the diagnosis of sepsis or other diseases was confirmed (≤ 7 days); 2) Follow-up period: after the diagnosis of sepsis, the subjects will be followed up for 28 days.
  Comparing to reference method, the clinical diagnosis of sepsis (sepsis-3), and reference reagents, CE-marked IVD PSP capsule on the point-of-care abioSCOPE® device (Abionic SA), C-reactive protein (CRP) assay kit, procalcitonin (PCT) assay kit, etc., to verify and evaluate the comprehensive performance of PSP as a biomarker in the early recognition and diagnosis of sepsis in Chinese patient population manifesting within the first 3 days after testing. Diagnostic accuracy analysis and consistency analysis will be performed.

SECONDARY OUTCOMES:
Diagnostic performance of "PSP+X" model to aid in the early recognition and diagnosis of sepsis manifesting within the first 3 days after testing | 1) Blood sample collection period: from enrollment to the diagnosis of sepsis or other diseases was confirmed (≤ 7 days); 2) Follow-up period: after the diagnosis of sepsis, the subjects will be followed up for 28 days.
  Comparing to the reference method and the reference reagent test results, try to use machine learning & deep learning methods to select a subset of relevant features (variable screening) from clinical information and biomarker data (CRP, PCT, IL-6, NT-proBNP, hs-cTnI, SAA, Cys C, CAL, etc.), to construct an innovative combined diagnostic model (named it "PSP+X" index) with PSP by logistic regression. The receiver operating characteristic curve (ROC) analysis is used to evaluate the diagnostic value of "PSP+X" index for the early recognition and diagnosis of sepsis manifesting within the first 3 days after testing will be evaluated.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong